CLINICAL TRIAL: NCT06237829
Title: Testing Tactile Aids With Blind Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 372362
Record Dates: First submitted 2023-11-30; First posted 2024-02-02 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Vision, Low; Blindness
Keywords: Tactile Aid
MeSH Terms: conditions — Vision, Low; Blindness

STUDY DESIGN:
Intervention Model Description: Groups of participants will proceed with tactile aids in increasingly higher levels of complexity. The primary evaluation of participant outcome is the success rate with which they can correctly distinguish between multiple surfaces. In the first intervention, participants will be asked to categorize two different coated materials into their respective categories by touch. Participants who score 65% or higher, will be asked to continue. In the second intervention, participants will be asked to categorize four different coated materials into their respective categories. Participants who statistically significantly above chance can identify coated materials successfully will be asked to continue. In the last intervention, participants will be asked to identify between multiple categories on a tactile chart made from a combination of traditional physical features denoting categories and the coatings under investigation denoting another category.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Identifying and synthesizing high-contrast tactile materials without physical features (Experimental): Beyond the few materials investigators previously identified, it is unknown which materials are useful for creating tactile sensations. Common material properties such as a friction coefficient or hydrophilicity are insufficiently detailed to accurately predict friction forces-the basis of tactile stimuli. The investigators will use expertise in connecting tactile sensations with chemical structure through mechanical testing, theory, and human testing. The investigators' goal is to identify materials that lead to high tactile contrast without relying on physical features. (Tactile contrast is defined by the investigators as large differences in friction which are easily distinguishable by humans during free tactile exploration.)
  Interventions: Behavioral: Single bump acuity; Behavioral: Optimal spacing between bumps; Behavioral: Improving signal from a single bump with designer materials
- Building tactile aids with designer materials for plots, games, and object labeling (Experimental): Investigators will build static tactile aids with designer materials, i.e., silanes and polymers coatings. These aids will be a mathematical plot, a board game, and simulated money. Investigators will compare the speed, accuracy, and amount of information of hybrid tactile aids made from designer materials and physical features to traditional tactile aids made only with bumps.
  Interventions: Behavioral: Single bump acuity; Behavioral: Optimal spacing between bumps; Behavioral: Improving signal from a single bump with designer materials
- Optimal design of bumps and designer materials in tactile aids (Experimental): Reflecting the lack of standardized methods or benchmarks for tactile technologies, the known limits of tactile sensitivity was narrowed from millimeters, microns, to nanometers within the last 10 years by use of metal wires, wrinkled plastics, and silanes, respectively. Investigators will determine the optimal design of traditional bumps which yields the highest tactile stimulus in the smallest area. Investigators expect to find that current bumps are larger than necessary, and that the same information could be placed into a smaller area (higher information density). Then, investigators will augment bumps with designer materials to increase the tactile stimulus from a bump, thereby permitting even smaller bumps to increase information density. Beyond optimal design methods, the investigators' quantitative methods, enabled by making the mechanical stimulus the dependent variable, also serve as benchmarks between tactile aids.
  Interventions: Behavioral: Single bump acuity; Behavioral: Optimal spacing between bumps; Behavioral: Improving signal from a single bump with designer materials

INTERVENTIONS:
Behavioral: Single bump acuity — Investigators will design bumps of varying heights, spacings, diameters, and bump shapes (rounded top, flat top, angled top) which give a precise amount of mechanical stimulus to the finger. Subjects will be asked if they could notice a bump on the surface and instructed to make the judgment quickly (<2 seconds). A psychometric curve, with a standard braille bump serving as the positive, ~100% success rate control, will be constructed
Behavioral: Optimal spacing between bumps — Investigators will fabricate and characterize two bumps of varying widths (ranging from 150 μm to 3 times the bump width, based on fabrication resolution available in commercial tactile aid machines). Subjects will be asked to run their finger across the two bumps (two bumps always form a line, so investigators do not need to ask subjects to orient their fingers) quickly and asked if they felt one bump or two.
Behavioral: Improving signal from a single bump with designer materials — Investigators will coat single bumps with our designer materials (with alkyl and amino functional groups) to improve the mechanical stimuli from a single bump. Subjects will then be asked to perform a similar experiment as the "single bump acuity" test and the "optimal spacing between bumps" test. ("can you notice the bump?" or "did you feel one or two bumps").

SUMMARY:
The objective of this project is to create richer tactile aids by using materials chemistry to create tactile sensations in tactile aids, as an alternative to traditional physical bumps, lines, or textures. These materials are commonly used in household products, but have not yet been used to enrich tactile aids. Successful outcomes are primarily the accuracy with which low vision or blind subjects identify objects made from tactile coatings versus traditional tactile aids. Other outcomes include time to completion of the task, or the number of distinctive categories that participants can identify.

DETAILED DESCRIPTION:
Traditional images and graphics, like mathematical plots or charts, are not accessible to low vision and blind people. Instead, for blind and low vision people, tactile aids are traditionally used to convey abstract concepts. However, tactile aids cannot convey as rich or as dense of information as traditional visual graphics, limiting independence and access to gainful employment for low vision and blind professionals.

The primary reason why tactile aids are inferior to visual graphics is that tactile aids are made from a combination of physical bumps, lines, and labels. Placing too many details on a single tactile aid quickly becomes illegible to the user because the various bumps, lines, and textures blur together, which is known as "tactile clutter".

The objective of this project is to create richer tactile aids by using materials chemistry to create tactile sensations in tactile aids, as an alternative to traditional physical bumps, lines, or textures. These materials are commonly used in household products, but have not yet been used to enrich tactile aids. Successful outcomes include having low vision or blind subjects identify objects made from our tactile materials quicker than traditional tactile aids, or to successfully identify more categories on a mathematical plot than is currently possible with existing tactile aids.

ELIGIBILITY:
Inclusion Criteria:

* Visual Impairment: Participants should be blind or visually impaired for greater than 10 years, either congenitally or acquired.
* Tactile Aid Usage: Participants must use tactile aids regularly.
* Mathematical Knowledge: Participants should have a basic understanding of mathematical plots, equivalent to at least high school geometry.

Exclusion Criteria:

- Limb Conditions: Participants with amputations or outer extremity conditions affecting hand use will be excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Success rate for correctly interpreting a tactile numeric plot of the GDP (Gross Domestic Product) of four countries. | Immediately after human testing (middle of year 2)
  Researchers will create a tactile plot of the GDP of four countries on an xy plot. The different countries are denoted from a combination of traditional lines or bump-dashed lines, and from a line made with a tactile coating. At three positions along the x-axis of on the plot, the relative GDP of which country has the most will change. Participants will be asked to give which country is the highest GDP and the lowest at these three positions. The primary outcome measure is if when asked, what is the GDP of country X at a certain value, participants successfully provide the correct value. More specifically, the percent of answer correct for each given country. Four countries will be used, with three being denoted through physical features, and the fourth denoted with a tactile coating.
Usability of GDP plot tactile aid. | Immediately after human testing (middle of year 2)
  Researchers will create a tactile plot of the GDP of four countries on an xy plot. The different countries are denoted from a combination of traditional lines or bump-dashed lines, and from a line made with a tactile coating. At three positions along the x-axis of on the plot, the relative GDP of which country has the most will change. Participants will be asked to give which country is the highest GDP and the lowest at these three positions. Secondary outcome measures are usability of the tactile aid on a Likert scale, its comfort, how easy the tactile coating was to distinguish versus the physical features, and a free response of feedback on usability.
  Title: GDP Plot Usability Min: 0 Max: 6 Higher the score, the better the outcome/ usability of the tactile plot.
Time to completion of a tactile board game. | Immediately after human testing with this tactile aid (end of year 3)
  For participants who were successful at the Outcome 1 Task, they will be asked to play a tactile board game that resembles "chutes and ladders". They will play one of two versions, with the first version being randomized across participants. In one version, the chutes and ladders are made from traditional physical features. In the second version, the chutes and ladder each have tactile coatings in addition to their physical features. Participants will be given a preselected list of spaces to move which normalizes the path length between the board made with only physical features versus the board made with physical features and tactile coatings. Participants will be timed on how quickly they finish the board game and the time to completion between the two different boards will be compared.
Success rate to completion for a fake money counting task. | Immediately after human testing with this tactile aid (end of year 4)
  Participants will be given a random collection of 3-5 fake bills with the denominations on the bills each represented by a different tactile coating. After familiarization and training, participants will be given the random collection of 3-5 fake bills and asked to give a sum of the bills in their hand. Participants will be evaluated on whether or not their response is correct. This will be repeated 15 times.
Success time to completion for a fake money counting task. | Immediately after human testing with this tactile aid (end of year 4)
  Participants will be given a random collection of 3-5 fake bills with the denominations on the bills each represented by a different tactile coating. After familiarization and training, participants will be given the random collection of 3-5 fake bills and asked to give a sum of the bills in their hand. Participants will be evaluated on how quickly they completed the task. This will be repeated 15 times.
Usability and general feedback | Through study completion, 4 years.
  Subjects participating in the clinical trial will be invited to provide feedback on the usability and their preferences regarding the tactile aid introduced in the study. The assessment will be conducted using a modified Likert scale. This outcome aims to gather subjective experiences related to the use of new tactile aids throughout the trials. Throughout the study, participants will be consistently asked to comment on the usability and their preferences based on the tactile aid. This ongoing feedback will enable a comprehensive understanding of their experiences over time.
  Modified Likert Scale:
  Strongly Disagree Disagree Somewhat Disagree Neutral Somewhat Agree Agree Strongly Agree Extremely Agree Exceptionally Agree
  Title: Usability of Tactile Aid Min: 1 Max: 9 Higher the score, the better the outcome/ usability of the tactile aid.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No